CLINICAL TRIAL: NCT00386204
Title: Efficacy and Side Effects of Q-Switched Ruby Laser Treatment of Solar Lentigines in Two Different Fitzpatrick Skin Types II and IV
Brief Title: Side Effects of Q-Switched Ruby Laser for the Treatment of Lentigines in Light and Dark Skin Types
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: src-pts-11073
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Solar Lentigines
Keywords: Q-switched Ruby laser

INTERVENTIONS:
Device: Q-switched Ruby Laser

SUMMARY:
The purpose of this study is a comparison of efficacy and side effects of Q-switched Ruby laser treatment for solar lentigines in two different skin types II and IV.

DETAILED DESCRIPTION:
It has been widely accepted that dark colored individuals are prone to develop laser induced side effects especially post inflammatory hyperpigmentation(PIH) and it could be a limiting issue in selecting dark colored individuals.

We designed this study to evaluate the difference of efficacy and side effects in light and dark skinned individuals.

ELIGIBILITY:
Inclusion Criteria:

* Solar Lentigines
* Fitzpatrick skin type II and IV

Exclusion Criteria:

* Pregnancy
* Age above 80
* Photosensitivity
* Concern for malignancy
* Active Infection

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2005-11; Study Completion 2006-09

PRIMARY OUTCOMES:
Clinical Clearance
Side Effects

CONTACTS AND LOCATIONS:
Overall Officials: Parviz Toossi, M.D., Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Skin Research Center, Shohada-e Tajrish Hospital, Shaheed Beheshti Medical University, Tehran, Tehran Province, Iran